CLINICAL TRIAL: NCT03811600
Title: Exosomes Implication in PD1-PD-L1 Pathway Activation in Obstructive Sleep Apnea Syndrome
Brief Title: Exosomes Implication in PD1-PD-L1 Activation in OSAS
Acronym: ExoSAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-A00029-48
Record Dates: First submitted 2019-01-15; First posted 2019-01-22 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-05

CONDITIONS: Sleep Apnea Syndromes, Obstructive; Cancer
MeSH Terms: conditions — Sleep Apnea Syndromes; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSAS patients: 45 patients investigated for suspected OSAS with an apnea hypopnea index ≥15 per hour
  Interventions: Diagnostic Test: PD1/PD-L1 exosomal expression
- Non OSAS patients: 45 patients investigated for suspected OSAS with an apnea hypopnea index <15 per hour
  Interventions: Diagnostic Test: PD1/PD-L1 exosomal expression

INTERVENTIONS:
Diagnostic Test: PD1/PD-L1 exosomal expression — exosomal PD1/PD-L1 expression

SUMMARY:
An increased occurrence of cancer associated mortality has been described in patients with Obstructive Sleep Apnea Syndrome (OSAS). This association might be partially explained by an impaired cellular immune response that has been described in OSAS. Is has been suggested that OSAS impact immune cells by upregulation of the PD-1/PD-L1 pathway. Exosomes are small membrane vesicles released by numerous cells in the bloodstream. Exosomes have been shown to be implicated in cancer cells proliferation via a PD-1/PD-L1 pathway activation.

This study will evaluate exosomal PD-1/PD-L1 expression in patients with OSAS as compared to controls and will further investigate their impact on immune cells function and proliferation capacities.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a sleep recording for suspected OSAS

Exclusion Criteria:

* Préviously treated OSAS
* Cancer past history
* Pregnant women
* Cognitif impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients investigated by sleep recording for suspected OSAS will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
exosomal PD1 expression | at baseline
  Peripheral blood (≈20 ml) will be collected from non-OSAS or OSAS subjects on EDTA-coated tubes. Exosomes will be isolated by centrifugation. For detecting exosome-associated surface proteins by flow cytometry, exosomes will be first captured on magnetic beads. The bead/exosome complexes will be then co-incubated with the labeled detection antibodies, either anti-PD1. Next, the complexes will be washed 3x resuspended in 300uL of PBS for antigen detection by flow cytometry.
exosomal PD-L1 expression | at baseline
  Peripheral blood (≈20 ml) will be collected from non-OSAS or OSAS subjects on EDTA-coated tubes. Exosomes will be isolated by centrifugation. For detecting exosome-associated surface proteins by flow cytometry, exosomes will be first captured on magnetic beads. The bead/exosome complexes will be then co-incubated with the labeled detection antibodies, either anti-PD-L1. Next, the complexes will be washed 3x resuspended in 300uL of PBS for antigen detection by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire du Sommeil, Département de Pneumologie, CHU d'Angers, Angers, France